CLINICAL TRIAL: NCT01165411
Title: Developing and Maintaining a Central Venous Catheter Registry
Status: Completed | Type: Observational
Sponsor: Lehigh Valley Hospital (Other)
Responsible Party: Principal Investigator, Marna Rayl Greenberg, Director of EM Research, Lehigh Valley Hospital
Other Study IDs: Registry
Record Dates: First submitted 2010-07-12; First posted 2010-07-19 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Infection
Keywords: Central Catheterization; Central Line; Database; Registry; Registries
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with CVCs and PICC lines placed: This group will have either Standard of Care (control) or Process Improvement infection control changes administered.

SUMMARY:
It has been estimated that 90% of bloodstream infections associated with catheters, are due to CVCs, and that 500 to 4,000 patients in the United States die annually due to these bloodstream infections. The risk of central line associated bloodstream infections is typically expressed as the number of line infections per 1000 catheter days. This study's goal is to develop a uniform CL protocol, updated practice guidelines based on current evidence, and a standard procedural checklist based on CL care bundles recommended by the Institute for Healthcare Improvement. A secondary goal is to create a CL registry to capture and store data relevant to each CL placed throughout the institution. This registry will provide a wealth of data on CL insertions and complications that may be used as a valuable source of information for quality assurance, performance improvement, and research. With the knowledge and information obtained through this registry, educational offerings can be created, and a standardized institutional process for CL insertion can be developed.

DETAILED DESCRIPTION:
The use of central venous catheters(CVCs) has increased in both the inpatient and outpatient settings.CVCs disturb skin integrity and create vulnerability for bacterial and fungal infections. It has been estimated that 90% of bloodstream infections associated with catheters, are due to CVCs, and that 500 to 4,000 patients in the United States die annually due to these bloodstream infections (Mermel, 2000). The risk of central line (CL)associated bloodstream infections (CLAB) is typically expressed as the number of line infections per 1000 catheter days.A recent study demonstrated that following a set of standardized procedures can reduce the mean CLAB rate from 7.7 per 1000 catheter days to 1.4 (Pronovost et al., 2006).In an effort to decrease hospital acquired bloodstream infections and complications resulting from CVCs, an initiative to standardize and track CL placement throughout the institution is proposed. A uniform CL protocol will be developed;practice guidelines will be updated based on current evidence, and a standard procedural checklist will be developed based on CL care bundles recommended by the Institute for Healthcare Improvement (IHI)(5 Million Lives, 2007).Generally,a care bundle is a series of best practices that each enhances care when applied individually, but considerably improves care when implemented together.The CL care bundle includes hand hygiene, barrier precautions, chlorhexidine skin antisepsis, optimal site selection, and daily consideration of line necessity, with timely removal of unnecessary lines(5 Million Lives, 2007).Another goal of this initiative is to create a CL registry to capture and store data relevant to each CL placed throughout the institution.This registry will provide a wealth of data on CL insertions and complications which may be used as a valuable source of information for quality assurance, performance improvement, and research.Finally,with the knowledge and information obtained through this registry, educational offerings can be created, and a standardized institutional process for CL insertion can be developed.

Objective: 1.To capture information on each CL insertion throughout the institution.2.To capture and track the amount of days a patient has a CL in place.3.To capture and track CL infectious complications.4.To capture and track mechanical complications.5.To capture data,which may be used as a valuable source of information for quality assurance, performance improvement, education, and research.

ELIGIBILITY:
Inclusion Criteria:

* All patients that have CVCs and PICC lines placed at LVH.

Exclusion Criteria:

* The patient has a CVC or PICC that was placed outside of LVHN.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients that have CVCs and PICC lines placed at LVH
Sampling Method: Non-Probability Sample
Enrollment: 4530 (Actual)
Dates: Start 2008-08; Primary Completion 2015-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Track and store data on central line insertions and complications which may be used as a valuable source of information for quality assurance, performance improvement, and research | At time of complication or infection
  All data elements collected are either part of the standard of care during routine insertion of Central Venous Catheters (CVCs) and Peripheral Inserted Central Catheter (PICCs) or are undergoing process improvement so that they become the standard of care for these lines.
  The hospital data warehouse will be automatically fed information from multiple existing databases that are maintained within different locations of the hospital. Once merged, data will be transferred into the Horizon Business Insight database for performance improvement, quality assurance, and research purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie A Rupp, RN, BSN, Principal Investigator — Lehigh Valley Health Network
Locations (1):
- Lehigh Valley Health Network, Allentown, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mermel LA. Prevention of intravascular catheter-related infections. Ann Intern Med. 2000 Mar 7;132(5):391-402. doi: 10.7326/0003-4819-132-5-200003070-00009. PMID 10691590
- [Background] DerGurahian J. 5 million lives campaign hits midway point . . . but Institute for Healthcare Improvement officials say it's hard to judge progress. Mod Healthc. 2007 Dec 17;37(50):12-3. No abstract available. PMID 18203368
- [Background] Pronovost P, Needham D, Berenholtz S, Sinopoli D, Chu H, Cosgrove S, Sexton B, Hyzy R, Welsh R, Roth G, Bander J, Kepros J, Goeschel C. An intervention to decrease catheter-related bloodstream infections in the ICU. N Engl J Med. 2006 Dec 28;355(26):2725-32. doi: 10.1056/NEJMoa061115. PMID 17192537